CLINICAL TRIAL: NCT02700204
Title: Histological Study to Evaluate Skin Changes After PicoWay® 1064 nm and 532nm Picosecond Fractional Laser Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DHF19921
Record Dates: First submitted 2016-02-28; First posted 2016-03-07 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Dyschromia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PicoWay 532nm fractional treatment (Experimental): subjects will receive one treatment for peri auricular and/or Buttocks by 532nm hand-piece
  Interventions: Device: PicoWay 532nm fractional treatment
- PicoWay 1064nm fractional treatment (Experimental): subjects will receive one treatment for peri auricular and/or Buttocks by 1064nm hand-piece
  Interventions: Device: PicoWay 1064nm fractional treatment

INTERVENTIONS:
Device: PicoWay 532nm fractional treatment — is a solid state laser capable of delivering energy at dual wavelength of 1064 nm or 532 nm at extremely short durations in the range of 300-900 ps
  Other Names: PicoWay Resolve 532nm handpiece
  Arms: PicoWay 532nm fractional treatment
Device: PicoWay 1064nm fractional treatment — is a solid state laser capable of delivering energy at dual wavelength of 1064 nm or 532 nm at extremely short durations in the range of 300-900 ps
  Other Names: PicoWay Resolve 1064nm handpiece
  Arms: PicoWay 1064nm fractional treatment

SUMMARY:
This is an open-label, two-arm, histological evaluation study.

Subjects in this study will be assigned to Arm 1 or Arm 2, taking into account skin type, to receive PicoWay fractional treatment:

Arm 1: 532nm hand-piece Arm 2: 1064nm hand-piece Subjects will receive one treatment for peri auricular and/or Buttocks according the Investigator decision, with the fractional hand-piece

All subjects will have biopsies from the treated area:

* at baseline prior to treatment;
* immediately after treatment (within 30 minutes) or 48 hours after treatment;
* 2 months after treatment. Methodology described in the protocol to evaluate efficacy and safety of treatments will be carried out at each visit at the clinic.

DETAILED DESCRIPTION:
This histological study is a prospective clinical study to evaluate skin biopsies after a single PicoWay treatment with the 532nm or 1064nm fractional hand-piece.

Up to 30 healthy candidates, will be enrolled at up to 2 participating study sites. Subjects in this study will be assigned to Arm 1 or Arm 2, taking into account skin type, to receive fractional treatment for peri auricular and/or Buttocks according to investigator decision:

Arm 1: 532nm hand-piece Arm 2: 1064nm hand-piece

Subjects will receive one treatment for peri auricular and/or Buttocks, with the fractional hand-piece. The investigator may use a multiplicity of energy levels in area or subarea in a single treatment, in order to titrate the optimum energy level. Further, if the investigator elects to, the Picoway handpiece can have at its distal end (at the distance gauge ending) a flat piece of a transparent plastic/glass (with appropriate anti reflective coating if desired), which will be in contact with the skin. In this case, the investigator may also elect to use a coupling gel as a matching medium between the skin and the glass.

All subjects will have biopsies of the treated area (a single or two peri or post-auricular, buttocks) at baseline prior to treatment. Biopsies from each area will also be performed immediately after treatment (within 30 minutes) and/or at ~48 hours after treatment, according to physician discretion, and at the 2-month follow-up.

Topical anesthetic (ointment) or intradermal injected solution may be used prior to treatment

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female and male subjects between 18 to 75 years of age
2. Has Fitzpatrick skin type I-VI
3. Subjects seeking treatment for having blemished skin, where the blemishes are of the type that photo rejuvenation would be a potential treatment option, including dyschromia, acne scars, wrinkles, etc., and willing to undergo laser treatment and skin biopsies pre-treatment, immediately after treatment, and at the 2-month follow-up
4. Willing to receive the proposed PicoWay fractional treatments and comply with all study (protocol) requirements including consenting to a minimum of 5 biopsies: at least 1 biopsy pretreatment, at least 2 biopsies immediately after treatment (at least 1 from each side), or at least 2 biopsies at 48 hours after treatment (at least 1 from each side) and at least 2 biopsies at 2 months after treatment (at least 1 from each side)
5. Willing to have photographs and images taken of the treated areas to be used in evaluations, publications and presentations (subject identity will be masked)
6. For female subjects: not pregnant or lactating and is either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence)
7. Informed consent process is completed and subject consent is signed

Exclusion Criteria:

1. Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breast feeding
2. Hypersensitivity to light exposure
3. Active sun tan in facial area for patient who will treat peri-auricular area.
4. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions, hidradenitis, or dermatitis of the treatment area prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course
5. Is taking medication(s) for which sunlight is a contraindication
6. Has a history of squamous cell carcinoma or melanoma
7. History of keloid scarring, abnormal wound healing and / or prone to bruising
8. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity), including collagen vascular disease or vasculitic disorders
9. Has used oral isotretinoin (Accutane®) within 12 months of initial treatment or plans on using during the course of the study. Note: Skin must regain its normal degree of moisture prior to treatment, e.g., lack of noticeable skin flaking, skin peeling and skin surface roughness.
10. A laser procedure, a peel or has used lightening creams that was performed in the area to be treated with the past six months
11. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications
12. Known allergy to lidocaine, tetracaine, Xylocaine or epinephrine
13. Subjects with pigmented lesions that are considered not acceptable by the study investigator or any condition that, in the investigator's opinion, would make it unsafe to treat.
14. As per the investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
To collect skin biopsies after fractional PicoWay treatments | day 0 up to 2 months
  To collect skin biopsies after fractional PicoWay treatments to evaluate depth and damage caused by laser induced optical breakdown (LIOB)

SECONDARY OUTCOMES:
Histological evidence of LIOBs and location of LIOBs | day 0 and at 48 hours
  Histological evidence of LIOBs and location of LIOBs (epidermis or dermis) immediately after treatment or at 48 hours after treatment, with either the 1064nm or 532nm picosecond fractional laser focused at the surface or sub-surface of the peri auricular and/or Buttocks area/s
Observation of erythema/edema after treatment | day 0 up to 2 months
  Observation of erythema/edema after treatment via clinical skin assessment
Histological evidence of an inflammatory response | at 48 hours
  Histological evidence of an inflammatory response in the dermis immediately after treatment or at 48 hours after treatment that should lead to production of new collagen and elastin
Histological evidence of new collagen growth | at 2 months
  Histological evidence of new collagen growth at 2 months after treatment with either a 1064nm or 532nm picosecond fractional laser treatment
Number of subjects with adverse events | day 0, up to 7 months
  The number, description, severity, intervention and outcome of any adverse events will be reported on adverse event forms

CONTACTS AND LOCATIONS:
Overall Officials: Arielle Kauvar, MD, Principal Investigator — NY Laser Skin Care
Locations (1):
- Arielle N. Kauvar,, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brightman L, Goldman MP, Taub AF. Sublative rejuvenation: experience with a new fractional radiofrequency system for skin rejuvenation and repair. J Drugs Dermatol. 2009 Nov;8(11 Suppl):s9-13. PMID 19916261